CLINICAL TRIAL: NCT01244425
Title: A Randomized, Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Fibrin Sealant VH S/D 500 S-apr (Tisseel) for Hemostasis in Subjects Undergoing Hepatic Resection
Brief Title: Fibrin Sealant VH S/D 500 S-apr in Hepatic Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550904; 2010-018480-42 (EudraCT Number)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Bleeding (Oozing) in Hepatic Resection
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive; Low Density Lipoprotein Receptor-Related Protein-1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS VH S/D 500 s-apr (Experimental): Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant. Hemostasis will be assessed at 4, 6, 8 and 10 minutes after application of the study treatment.
  Interventions: Drug: Fibrin Sealant (FS) VH S/D 500 s-apr
- Manual compression - Control (Active Comparator): A dry surgical gauze swab will be used to apply by hand an even light pressure onto the oozing resection surface of the liver. Hemostasis will be assessed at 4, 6, 8 and 10 minutes after application of the study treatment.
  Interventions: Other: Manual compression

INTERVENTIONS:
Drug: Fibrin Sealant (FS) VH S/D 500 s-apr — Dosage form: spray application; dosage frequency: single application
  Other Names: Tisseel
  Arms: FS VH S/D 500 s-apr
Other: Manual compression — Dosage form: surgical gauze swab; dosage frequency: single application
  Arms: Manual compression - Control

SUMMARY:
The purpose of the study is to compare safety and efficacy of Fibrin Sealant (FS) Vapor Heated (VH) S/D 500 s-apr with manual compression as a supportive treatment of local bleeding (i.e. oozing) in hepatic resection surgery when standard surgical techniques are insufficient.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

* Signed informed consent obtained from the subject before any study-related activities
* Subject's age is 18 years or above
* Subject will undergo planned, elective resection of at least 1 anatomical segment of the liver for any reason by laparotomy
* Subject is willing and able to comply with the requirements of the protocol
* Female subjects of childbearing potential must present with a negative serum or urine pregnancy test within 72 hours before the elective liver resection
* Female subjects of childbearing potential must agree to employ adequate birth control measures for the time of their participation in the study

Intra-Operative Inclusion Criteria (before randomization):

* Resection of at least 1 anatomical segment of the liver has been performed
* Oozing from the cut surface of the liver persists after conventional resection procedure and primary control of arterial and venous bleeding by sutures, ligations, clips, vascular stapler, point electrocautery or focal radiofrequency ablation
* Need for additional supportive hemostatic treatment to stop bleeding (i.e. diffuse oozing) of the liver resection area

Pre-Operative Exclusion Criteria:

* Subject needs emergency liver surgery
* Subject will undergo liver resection via laparoscopic procedure
* Subject has known congenital coagulation disorder (e.g. hemophilia)
* Subject has known hypersensitivity to any ingredient of the investigational medicinal product
* Suspected inability or unwillingness of the subject to comply with trial procedures
* If female, subject is pregnant or lactating at the time of study enrollment
* Subject has already participated in this study (each subject can only be enrolled once)
* Subject has participated in another clinical study involving an investigational product or investigational device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an investigational product or investigational device during the course of this study

Intra-operative Exclusion Criteria (before randomization):

* Occurrence of any severe surgical complication that require resuscitation or deviation from the planned surgical procedure
* Disseminated intravascular coagulopathy (DIC)
* Application of any topical hemostatic material on the resection surface of the liver prior to application of the study treatment
* Radiofrequency precoagulation of the liver resection surface, except focal use of radiofrequency as primary hemostatic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Medical Director, MD, Study Director — Baxter Healthcare Corporation
Locations (7):
- Germany (7):
  - Berlin
  - Essen
  - Hanover
  - Heidelberg
  - Jena
  - Leipzig
  - Tübingen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 95 participants were enrolled and screened. 23 were screen failures. 2 participants were discontinued due to: 1 was operated on by a surgeon other than the investigator, and the other underwent a prolonged operation- meaning that the investigational product (IP) could not be used. Therefore, 70 of the 95 enrolled were randomized.
Period: Overall Study
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Started | 35 | 35
Completed | 32 (Adverse Event: multi-organ failure (death)) | 32 (Adverse Event: septic shock with multi-organ failure due to liver abscess (death))
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control | Total
Number analyzed (Participants) | 35 | 35 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (14.5) | 59.8 (12.8) | 57.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  Germany | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Intraoperative Hemostasis at 4 Minutes After Treatment Application
Description: Hemostasis defined as no visible bleeding on the liver resection surface (liver surgical site) after treatment application. Hemostasis had to be maintained until surgical closure. Time recording started with treatment application, ie, with the start of spraying Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) or with the application of manual compression.
  The following were regarded as treatment failures:
  * No hemostasis achieved at 4 minutes post treatment application (for the FS VH S/D 500 s-apr arm, the "time to hemostasis" was used; a time window of +5 seconds was acceptable for showing a success)
  * Additional hemostatic treatment (ie, hemostatics in addition to the randomized treatment) was required
  * Reapplication of FS VH S/D 500 s-apr after 4 minutes
  * Intraoperative rebleeding after the first 4 minutes of the observation period
Time Frame: 4 minutes post start of treatment application
Population: full analysis (data) set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant. Hemostasis will be assessed at 4 minutes after application of the study treatment.
- Manual Compression - Control: A dry surgical gauze swab will be used to apply by hand an even light pressure onto the resection surface of the liver. Hemostasis will be assessed at 4 minutes after application of the study treatment.
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 82.9 [68.3 to 92.8] | 37.1 [22.5 to 53.6]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p < 0.001, likelihood-ratio chi square test

2. Secondary Outcome: Percentage of Participants With Intraoperative Hemostasis at 6 Minutes After Application of the Randomized Treatment
Description: Hemostasis defined as no visible bleeding on the liver resection surface (liver surgical site) after treatment application. Hemostasis had to be maintained until surgical closure. Time recording started with treatment application, ie, with the start of spraying Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) or with the application of manual compression.
Time Frame: 6 minutes after start of treatment application
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant. Hemostasis will be assessed at 6 minutes after application of the study treatment.
- Manual Compression - Control: A dry surgical gauze swab will be used to apply by hand an even light pressure onto the resection surface of the liver. Hemostasis will be assessed at 6 minutes after application of the study treatment.
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 91.4 [79.3 to 97.8] | 57.1 [40.7 to 72.6]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p < 0.001, likelihood ratio chi-square test

3. Secondary Outcome: Percentage of Participants With Intraoperative Hemostasis at 8 Minutes After Application of the Randomized Treatment
Description: as for outcome 2
Time Frame: 8 minutes after start of treatment application
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant. Hemostasis will be assessed at 8 minutes after application of the study treatment.
- Manual Compression - Control: A dry surgical gauze swab will be used to apply by hand an even light pressure onto the resection surface of the liver. Hemostasis will be assessed at 8 minutes after application of the study treatment.
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 91.4 [79.3 to 97.8] | 71.4 [55.3 to 84.5]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p = 0.028, likelihood ratio chi-square test

4. Secondary Outcome: Percentage of Participants With Intraoperative Hemostasis at 10 Minutes After Application of the Randomized Treatment
Description: as for outcome 2
Time Frame: 10 minutes after start of treatment application
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant. Hemostasis will be assessed at 10 minutes after application of the study treatment.
- Manual Compression - Control: A dry surgical gauze swab will be used to apply by hand an even light pressure onto the resection surface of the liver. Hemostasis will be assessed at 10 minutes after application of the study treatment.
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 94.3 [83.4 to 99.0] | 74.3 [58.4 to 86.7]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p = 0.017, likelihood ratio chi-square test

5. Secondary Outcome: Percentage of Participants With Intraoperative Rebleeding After Occurrence of Hemostasis
Description: Intraoperative rebleeding from the treated liver resection surface after occurrence of hemostasis.
Time Frame: Intraoperative day 0
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Fibrin Sealant, Vapor Heated, Solvent/Detergent treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), not to exceed 20mL per participant.
- Manual Compression - Control: A dry surgical gauze swab will be used to apply by hand an even light pressure onto the resection surface of the liver.
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 2.9 [0.2 to 12.0] | 8.6 [2.2 to 20.7]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p = 0.293, likelihood ratio chi-square test

6. Secondary Outcome: Percentage of Participants With Postoperative Rebleeding
Description: Rebleeding until discharged from the surgical ward, defined as any rebleeding from the treated liver resection surface requiring surgical reexploration
Time Frame: Postoperative until discharged from surgical ward
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
Percentage of participants | 2.9 [0.1 to 14.9] | 0.0 [0.0 to 10.0]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p = 0.237, likelihood ratio chi-square test

7. Secondary Outcome: Percentage of Participants With Transfusion Requirements Until Discharged From Surgical Ward
Description: Transfusions administered included whole blood, packed red blood cells, fresh frozen plasma, and thrombocyte concentrate.
Time Frame: Intra- and postoperative until discharged from surgical ward
Population: Full analysis (data) set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 35 | 35
percentage of participants | 40.0 [24.9 to 56.5] | 42.9 [27.4 to 59.3]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Manual Compression - Control; Test type: Superiority or Other; p = 0.808, likelihood ratio chi-square test

8. Secondary Outcome: Median Total Volume of Postoperative Drainage Fluid Within 48 Hours After Surgery
Time Frame: Within 48 hours after surgery
Population: * Full analysis (data) set
  * Participants who received a drain and for whom the volume for the first 48 hours after surgery is available
Measure: Median (Full Range); unit: mL
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Number analyzed (Participants) | 32 | 31
mL | 415.0 [70 to 10800] | 410.0 [0 to 3690]

ADVERSE EVENTS:
Time Frame: Throughout study period (9 months)
Arm/Group | FS VH S/D 500 S-apr | Manual Compression - Control
Serious Adverse Events (participants affected / at risk) | 9/35 | 11/35
Other Adverse Events (participants affected / at risk) | 22/35 | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS VH S/D 500 S-apr (N=35) | Manual Compression - Control (N=35)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 2 (2)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 3 (3)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SUBDIAPHRAGMATIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SMALL-FOR-SIZE LIVER SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS VH S/D 500 S-apr (N=35) | Manual Compression - Control (N=35)
ASCITES (Gastrointestinal disorders) | 1 (1) | 4 (4)
IMPAIRED HEALING (General disorders) | 1 (1) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 2 (2)
INFECTION (Infections and infestations) | 2 (2) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
CHEMICAL PERITONITIS (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (14)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (3) | 2 (2)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)